CLINICAL TRIAL: NCT00504699
Title: Safety of Ovarian Stimulation With Letrozole and Gonadotropins in Breast Cancer Patients Undergoing Embryo or Oocyte Cryopreservation: A Prospective Controlled Follow up Study
Brief Title: Safety of Ovarian Stimulation With Letrozole and Gonadotropins in Breast Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI left the Institution.
Sponsor: New York Medical College (Other)
Responsible Party: Principal Investigator, kutluk oktay, PI, New York Medical College
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0110005172
Record Dates: First submitted 2007-07-18; First posted 2007-07-20 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer
Keywords: breast cancer; ovarian stimulation; aromatase inhibitors; letrozole; fertility preservation; recurrence
MeSH Terms: conditions — Breast Neoplasms; Recurrence | interventions — Ovulation Induction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- letrozole (Experimental): ovarian stimulation after breast cancer diagnosis and before breast cancer treatment
  Interventions: Procedure: Ovarian stimulation in vitro fertilization cryopreservation
- control (No Intervention): No ovarian stimulation before breast cancer treatment

INTERVENTIONS:
Procedure: Ovarian stimulation in vitro fertilization cryopreservation — Letrozole 5 mg/day during ovarian stimulation
  Arms: letrozole

SUMMARY:
Breast cancer patients are commonly treated with drugs that eggs present in the ovary and may reduce their chance for getting pregnant. Their fertility can be preserved by stimulating their ovaries, collecting multiple eggs, fertilize them in the lab and freeze them. Ovarian stimulation increase their estrogen levels in blood.this may stimulate their cancer and increase chance for recurrence. If a medicine that prevent estrogen rise is used (letrozole), this may increase the safety of stimulation. In this study we compared ovarian stimulation in breast cancer patients using letrozole with those who did not undergo stimulation and showed that there is no increase risk for recurrence after a median follow up of 2 years

DETAILED DESCRIPTION:
215 women with breast cancer were evaluated for fertility preservation before chemotherapy. Of those, 79 elected to undergo controlled ovarian stimulation (COH) with letrozole and gonadotropins for embryo or oocyte cryopreservation. The 136 patients who declined served as controls.There were no significant differences between the study and control groups regarding age at diagnosis, breast cancer prognostic parameters (tumor size, grade, number of positive lymph nodes, estrogen receptor status, her2-neu overexpression and vascular space invasion), and chemotherapy regimens. There was no difference between the two groups in the projected 10 year relapse, breast cancer specific mortality or overall mortality. There were 3 recurrences or contralateral breast cancers (2 distant, 1 locoregional) in the letrozole group, and 11 in the control group (9 distant, 1 locoregional, 1 contralateral breast).

Comparison; breast cancer patients that underwent ovarian stimulation with letrozole+gonadotropins and those who declined ovarian stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years
* Biopsy proven breast cancer
* No prior chemotherapy or oophorectomy
* Regular menstrual cycles
* Normal basal FSH and estradiol

Exclusion Criteria:

* Stage 4 breast cancer

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2002-01; Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Breast cancer relapse free survival after ovarian stimulation | after chemotherapy to end of follow up

SECONDARY OUTCOMES:
Estradiol level, number of embryos cryopreserved, clinical pregnancy rate, ovarian reserve after chemotherapy | during stimulation, after stimulation and 1-2 years after chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Kutluk H Oktay, MD, FACOG, Principal Investigator — IFP
Locations (1):
- IFPn, Valhalla, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oktay K, Turan V, Bedoschi G, Pacheco FS, Moy F. Fertility Preservation Success Subsequent to Concurrent Aromatase Inhibitor Treatment and Ovarian Stimulation in Women With Breast Cancer. J Clin Oncol. 2015 Aug 1;33(22):2424-9. doi: 10.1200/JCO.2014.59.3723. Epub 2015 Jun 22. PMID 26101247
- [Derived] Reddy J, Turan V, Bedoschi G, Moy F, Oktay K. Triggering final oocyte maturation with gonadotropin-releasing hormone agonist (GnRHa) versus human chorionic gonadotropin (hCG) in breast cancer patients undergoing fertility preservation: an extended experience. J Assist Reprod Genet. 2014 Jul;31(7):927-32. doi: 10.1007/s10815-014-0248-6. Epub 2014 May 23. PMID 24854484
- [Derived] Azim AA, Costantini-Ferrando M, Oktay K. Safety of fertility preservation by ovarian stimulation with letrozole and gonadotropins in patients with breast cancer: a prospective controlled study. J Clin Oncol. 2008 Jun 1;26(16):2630-5. doi: 10.1200/JCO.2007.14.8700. PMID 18509175